CLINICAL TRIAL: NCT03085745
Title: Corticomotor Plasticity as a Biomarker for Functional Improvement After Botulinium Treatment in Writer's Cramp
Brief Title: Sensorimotor Mapping in Patients With Writer's Cramp
Acronym: IWCToxin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IWCToxin
Record Dates: First submitted 2017-02-24; First posted 2017-03-21 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Writer's Cramp
Keywords: Writer's cramp; Sensorimotor plasticity; TMS; Afferent inhibition; Motor mapping; Sensory mapping; adaptive sensorimotor synergies; fine motor control
MeSH Terms: conditions — Dystonic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Magnetic Stimulation (TMS) (Experimental): 15 patients suffering from a writer's cramp, aged 20-80 who are currently treated with botulinum toxin will receive single pulse TMS
  Interventions: Other: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation (TMS) — TMS is a non invasive brain stimulation technique which allows to measure corticospinal excitability from peripheral muscles.

SUMMARY:
Writer's cramp (WC) is a form of focal dystonia, a movement disorder characterized by sustained or intermittent muscle contractions causing abnormal, often repetitive movements, postures, or both. It typically manifests while writing, making handwriting impossible in the most severe cases. Treatment can be difficult, but one effective and well-tolerated treatment consists in local muscle injections with botulinum toxin. Although clinical improvement seems to be related to focal muscle chemodenervation, central plasticity changes may occur. The main aim of the study is to characterize and quantify the changes in intrinsic hand muscle cortical representations at rest and during isometric contractions of the finger muscles before and after treatment with botulinum toxin and the changes in sensorimotor integration in patients with writer's cramp.

DETAILED DESCRIPTION:
Fifteen WC patients will be enrolled in the study. A newly developed neuronavigated and robotized Transcranial Magnetic Stimulation (TMS) mapping approach will be used. It will generate a linear mediolateral excitability profile for two intrinsic hand muscle based on the mean Motor Evoked Potentials (MEPs) amplitude at each stimulation site. Changes in excitability profiles will reflect spatial reorganization of cortical motor output maps of the hand muscles. To measure afferent inhibition, the same mapping procedure will be repeated with a brief peripheral electrical stimulation prior the TMS pulse. These Short Afferent Inhibition (SAI) profiles will reflect the influence of the primary sensory cortex over the motor cortex. Finally, the stimulation grid will be translated to the primary somatosensory cortex and a paired pulse TMS paradigm will be applied just after a digital nerve stimulation. It will generate afferent signal processing profiles based on subjective perception for the index finger and the little finger. Participants will be tested before the botulinum toxin injections and at three different time points after the injections (7 days, 1 month and 3 months after). Botulinum toxin injections will be performed using ultrasound guide together with electromyography/nerve stimulation into the clinical affected hand muscles. Muscle selection for injections will be based on clinical criteria of postural deviation of the hand and fingers and responsible muscle forces. The dose will be chosen according to published clinical recommendation concerning starting dose for WC after the clinical examination, usually between 5 and 10 units of Xeomin® both for flexor and extensor hand/forearm muscles.

To precisely assess treatment efficacy, the Writer's Cramp Rating Scale (WCRS) as well as computer-based hand writing analyses and standard sensorimotor tests of hand functions (the Nine Holes Peg Test, a tapping test and a tactile spatial acuity task) will be performed before the injections and at each follow up session.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from a writer's cramp
* aged 30-80 years old
* Botulinum toxin injection performed in clinical routine for their disease
* Affiliated to a social security system
* Sufficient intellectual capacities to understand the tasks to perform
* Written consent obtained

Exclusion Criteria:

* Impossibility to remain sitting down without pain or discomfort for at least 3 consecutive hours
* History or psychiatric or neurological disease, different from dystonia.
* Subject under judicial oversight
* Subject being within exclusion period
* Subject not reachable in case of emergency,
* Presence of one or several contraindications to TMS
* Subject covered by the following articles from the french Code de la Santé Publique: L1121-5, L1121-6, L1121-7 et L1121-8.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-02-19 (Estimated); Study Completion 2019-05-19 (Estimated)

PRIMARY OUTCOMES:
Corticospinal excitability profiles of intrinsic hand muscles | This measure will be performed before the injection of botulinum toxin and 7 days after, 30 days after and 3 months after the injection.
  We will use a newly developed neuronavigated and robotized Transcranial Magnetic Stimulation (TMS) mapping approach consisting in an individually adjusted stimulation grid located along the longitudinal axis of the motor cortex. It will generate a linear mediolateral excitability profile for each hand muscle based on the mean Motor Evoked Potentials (MEPs) amplitude at each stimulation site, on both hemispheres. Changes in excitability profiles will reflect spatial reorganization of cortical motor output maps of the hand muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Elena MORO, Pr, Principal Investigator — amoro@chu-grenoble.fr
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided